CLINICAL TRIAL: NCT04036149
Title: Prospective Clinical Trial to Compare the Postoperative Horizontal Position Stability of the CT LUCIA 611P and the CT ASPHINA 409MP
Brief Title: To Compare Postoperative Horizontal Position Stability of the CT LUCIA 611P and the CT ASPHINA 409MP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT LUCIA 611P BER-401-16
Record Dates: First submitted 2019-07-26; First posted 2019-07-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Cataract Senile
MeSH Terms: interventions — Lenses, Intraocular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUCIA (Experimental): CT LUCIA 611P - Intraocular lens
  Interventions: Device: Intraocular lens
- ASPHINA (Active Comparator): CT ASPHINA 409MP - Intraocular lens
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Implantation as part of cataract surgery

SUMMARY:
The main objective of the trial is to assess the efficacy of the CT LUCIA 611P intraocular lens (IOL) with regard to the horizontal IOL position stability. The horizontal position collected at 1 month and 4 to 6 months post-operatively will be compared to the horizontal IOL position recorded at baseline (1 week post-operatively) as well as to the position stability of the reference IOL, CT ASPHINA 409MP.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent;
* Patients of any gender, aged 50 to 90 years;
* Assured follow-up examinations;
* Healthy eyes besides clinically significant bilateral age-related cataract.
* Distance corrected visual acuity ≤ 0.3 logMAR Normal findings in the medical history and physical examination
* Calculated IOL power within the available dioptre range;
* Biometry measurement/cataract density compatible with the IOLMaster evaluation.

Per operative inclusion criteria:

* IOL implanted in the capsular bag;
* The 2 IOL models (CT LUCIA 611P and CT ASPHINA 409MP) have been implanted in the 2 eyes of one patient;
* No intraoperative complications; no damaged capsular bag, no intraocular haemorrhage; no can opener rhexis.

Exclusion Criteria:

* Allergy to heparin
* Monophthalmic patient
* Ocular disorders, other than cataract, that could potentially cause future acuity loss to a level of 0.20 logMAR (best-corrected) or worse in either eye;
* Any anterior segment pathology that could significantly affect outcomes (e.g. chronic uveitis, iritis, corneal dystrophy, etc.);
* Floppy iris syndrome;
* Diabetic retinopathy;
* Traumatic cataract;
* Aniridia;
* Microphthalmus;
* Amblyopia;
* Degenerative visual disorders (e.g. macular degeneration, optic nerve atrophy, or retinal disorders);
* Patient expected to require retinal laser treatment before the end of the last follow-up;
* Previous intraocular and corneal surgery;
* Expected postop. astigmatism greater than 1 D;
* Any type of corneal disorder;
* Dementia;
* Pseudoexfoliation syndrome (PEX);
* Glaucoma or IOP higher than 24mmHg under ocular hypertension treatment;
* Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient.
* Pregnancy and/or lactation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Horizontal position stability | 1 week to 4-6 months post-operatively
  Evaluation of the horizontal position stability of the CT LUCIA 611P IOL. The horizontal position at M1 and M4-6 will be compared to the horizontal IOL position at baseline (W1) and to the position stability of the reference IOL, CT ASPHINA 409MP.

CONTACTS AND LOCATIONS:
Locations (1):
- VIROS, Hanusch Hospital, Department of Ophthalmology, Vienna, Austria